CLINICAL TRIAL: NCT05427721
Title: Thymol Administration Effects on Netrin-1 Serum Concentration on Obese Patients
Brief Title: Thymol on Netrin-1 on Obese Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Maria Guadalupe Ramos Zavala, Clinical Professor, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CI-01621; 20-131 (Registry Identifier: Research Coordination)
Record Dates: First submitted 2021-06-11; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Response; Obesity
Keywords: Netrin-1; Thymol
MeSH Terms: conditions — Obesity | interventions — Thymol

STUDY DESIGN:
Intervention Model Description: Clinical trial
Who Masked: Participant, Investigator
Masking Description: Capsules with the same characteristics (smell, color, taste). Random assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Thymol
  Interventions: Drug: Thymol
- Group B (Placebo Comparator): Calcined magnesia
  Interventions: Drug: Thymol

INTERVENTIONS:
Drug: Thymol — 200 mg each 8 hours for 90 days

SUMMARY:
The prevalence of obesity in Mexico is 35.4%, and it is considered a risk factor for the development of diabetes, systemic arterial hypertension and dyslipidemia. Obesity due to the increased distribution and growth of adipose tissue creates a pro-inflammatory state induced by molecules secreted by the adipocytes themselves. Netrin-1 is a cell migration protein, which directs the recruitment, migration and entrapment of macrophages in different tissues, within adipose tissue the entrapment of macrophages induces the release of pro-inflammatory cytokines, which increase the secretion of pro-inflammatory adipokines. It has been found in high concentration in patients with obesity, insulin resistance and type 2 diabetes. Thymol is a phytopharmaceutical derived from oregano oil that has shown powerful anti-inflammatory and antioxidant effects through the stimulation of PPAR-gamma, adiponectin and inhibition of the NF-κB pathway mediated by the JNK pathway, pathways in which netrin-1 is involved in macrophage entrapment and recruitment.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of thymol administration on the serum concentration of netrin-1 in obese subjects.

Material and methods: this is a randomized, double-blind, placebo-controlled clinical trial design.

Inclusion criteria:

1. - Subjects between 18 and 35 years old.
2. - Subjects with BMI ≥ 30.0 and ≤35.0.
3. - Subjects with systolic blood pressure less than 135 mmHg.
4. - Subjects with diastolic blood pressure less than 85 mmHg.
5. - Voluntary acceptance and signing of the informed consent. These patients will be randomly assigned to two groups, one will have the intervention with thymol 200 mg every 8 hours for 90 days while the other will have placebo with Mg 200 mg every 8 hours for 90 days.

Statistical analysis: quantitative variables: means and standard deviation. Qualitative variables: frequencies and percentages. In the comparison according to the serum level of netrin-1 between the two groups after the intervention: t student for quantitative variables, Chi square for qualitative variables. Statistical significance p equal to or less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 35 years old.
* BMI ≥ 30.0 and ≤35.0
* Systolic blood pressure less than 135 mmHg.
* Diastolic blood pressure less than 85 mmHg.

Exclusion Criteria:

* Subjects who are known to have a diagnosis, receive treatment, or are observed with:

  * Rheumatological and / or thyroid disease.
  * Chronic kidney disease and / or CKD-EPI glomerular filtration rate less than 60 ml / min / 1.72m2.
  * Innate alterations of metabolism.
  * Elevation of transaminases 2 times higher than normal.
  * Total cholesterol greater than 250 mg / dl.
  * Triglycerides greater than 300 mg / dl.
* Subjects presenting with acute illness, hospitalization, or drug treatment presented in the last 12 weeks prior to the study selection visit.
* Subjects with symptoms consistent with the definition of a probable case of COVID-19, as well as any subject with a diagnosis of COVID-19.
* Subjects who have had blood transfusions in the last 3 months.
* Regular smokers.
* Pregnant or lactating women.
* Women with a desire for pregnancy or who do not have a double barrier or progestin-only contraceptive method.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Netrin-1 | Change from baseline netrin-1 at 90 days
  Enzyme-Linked ImmunoSorbent Assay

SECONDARY OUTCOMES:
IL-6 | Change from baseline IL-6 at 90 days
  Enzyme-Linked ImmunoSorbent Assay
Adiponectin | Change from baseline adiponectin at 90 days
  Enzyme-Linked ImmunoSorbent Assay
Ultrasensitive C-reactive protein | Change from baseline hs-PCR at 90 days
  Enzyme-Linked ImmunoSorbent Assay

OTHER OUTCOMES:
Glucose | Change from baseline glucosa at 90 days
  Colorimetry
Insulin Insulina | Change from baseline insulina at 90 days
  Colorimetry
HDL | Change from baseline HDL at 90 days
  Colorimetry
LDL | Change from baseline LDL at 90 days
  Colorimetry
% visceral fat | Change from baseline % visceral fat at 90 days
  Bioelectrical impedance analysis
Abdominal Circumference | Change from baseline abdominal circumference at 90 days
  Centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Ramos-Zavala, PhD, Study Chair — Centro Universitario de Ciencias de la Salud, Mexico
Locations (1):
- INTEC, CUCS, Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammarstedt A, Gogg S, Hedjazifar S, Nerstedt A, Smith U. Impaired Adipogenesis and Dysfunctional Adipose Tissue in Human Hypertrophic Obesity. Physiol Rev. 2018 Oct 1;98(4):1911-1941. doi: 10.1152/physrev.00034.2017. PMID 30067159
- [Background] Stern JH, Rutkowski JM, Scherer PE. Adiponectin, Leptin, and Fatty Acids in the Maintenance of Metabolic Homeostasis through Adipose Tissue Crosstalk. Cell Metab. 2016 May 10;23(5):770-84. doi: 10.1016/j.cmet.2016.04.011. PMID 27166942
- [Background] Trayhurn P. Hypoxia and adipose tissue function and dysfunction in obesity. Physiol Rev. 2013 Jan;93(1):1-21. doi: 10.1152/physrev.00017.2012. PMID 23303904
- [Background] Han MS, Jung DY, Morel C, Lakhani SA, Kim JK, Flavell RA, Davis RJ. JNK expression by macrophages promotes obesity-induced insulin resistance and inflammation. Science. 2013 Jan 11;339(6116):218-22. doi: 10.1126/science.1227568. Epub 2012 Dec 6. PMID 23223452
- [Background] Lee KY, Gesta S, Boucher J, Wang XL, Kahn CR. The differential role of Hif1beta/Arnt and the hypoxic response in adipose function, fibrosis, and inflammation. Cell Metab. 2011 Oct 5;14(4):491-503. doi: 10.1016/j.cmet.2011.08.006. PMID 21982709
- [Background] Bouhlel MA, Derudas B, Rigamonti E, Dievart R, Brozek J, Haulon S, Zawadzki C, Jude B, Torpier G, Marx N, Staels B, Chinetti-Gbaguidi G. PPARgamma activation primes human monocytes into alternative M2 macrophages with anti-inflammatory properties. Cell Metab. 2007 Aug;6(2):137-43. doi: 10.1016/j.cmet.2007.06.010. PMID 17681149
- [Background] Yim J, Kim G, Lee BW, Kang ES, Cha BS, Kim JH, Cho JW, Lee SG, Lee YH. Relationship Between Circulating Netrin-1 Concentration, Impaired Fasting Glucose, and Newly Diagnosed Type 2 Diabetes. Front Endocrinol (Lausanne). 2018 Nov 23;9:691. doi: 10.3389/fendo.2018.00691. eCollection 2018. PMID 30532735
- [Background] Nagoor Meeran MF, Javed H, Al Taee H, Azimullah S, Ojha SK. Pharmacological Properties and Molecular Mechanisms of Thymol: Prospects for Its Therapeutic Potential and Pharmaceutical Development. Front Pharmacol. 2017 Jun 26;8:380. doi: 10.3389/fphar.2017.00380. eCollection 2017. PMID 28694777
- [Background] Nieddu M, Rassu G, Boatto G, Bosi P, Trevisi P, Giunchedi P, Carta A, Gavini E. Improvement of thymol properties by complexation with cyclodextrins: in vitro and in vivo studies. Carbohydr Polym. 2014 Feb 15;102:393-9. doi: 10.1016/j.carbpol.2013.10.084. Epub 2013 Nov 20. PMID 24507296
- [Background] Yu YM, Chao TY, Chang WC, Chang MJ, Lee MF. Thymol reduces oxidative stress, aortic intimal thickening, and inflammation-related gene expression in hyperlipidemic rabbits. J Food Drug Anal. 2016 Jul;24(3):556-563. doi: 10.1016/j.jfda.2016.02.004. Epub 2016 Apr 12. PMID 28911561
- [Background] Kohlert C, Schindler G, Marz RW, Abel G, Brinkhaus B, Derendorf H, Grafe EU, Veit M. Systemic availability and pharmacokinetics of thymol in humans. J Clin Pharmacol. 2002 Jul;42(7):731-7. doi: 10.1177/009127002401102678. PMID 12092740
- [Background] Salehi B, Mishra AP, Shukla I, Sharifi-Rad M, Contreras MDM, Segura-Carretero A, Fathi H, Nasrabadi NN, Kobarfard F, Sharifi-Rad J. Thymol, thyme, and other plant sources: Health and potential uses. Phytother Res. 2018 Sep;32(9):1688-1706. doi: 10.1002/ptr.6109. Epub 2018 May 22. PMID 29785774
- [Background] Paul S, Baranya Shrikrishna S, Suman E, Shenoy R, Rao A. Effect of fluoride varnish and chlorhexidine-thymol varnish on mutans streptococci levels in human dental plaque: a double-blinded randomized controlled trial. Int J Paediatr Dent. 2014 Nov;24(6):399-408. doi: 10.1111/ipd.12085. Epub 2013 Dec 25. PMID 24372823
- [Background] Marzouk T, Barakat R, Ragab A, Badria F, Badawy A. Lavender-thymol as a new topical aromatherapy preparation for episiotomy: A randomised clinical trial. J Obstet Gynaecol. 2015;35(5):472-5. doi: 10.3109/01443615.2014.970522. PMID 25384116 (Retraction: PMID 36350922 J Obstet Gynaecol. 2022 Nov 9;:1)
- [Background] Saravanan S, Pari L. Role of thymol on hyperglycemia and hyperlipidemia in high fat diet-induced type 2 diabetic C57BL/6J mice. Eur J Pharmacol. 2015 Aug 15;761:279-87. doi: 10.1016/j.ejphar.2015.05.034. Epub 2015 May 22. PMID 26007642
- [Background] Saravanan S, Pari L. Protective effect of thymol on high fat diet induced diabetic nephropathy in C57BL/6J mice. Chem Biol Interact. 2016 Feb 5;245:1-11. doi: 10.1016/j.cbi.2015.11.033. Epub 2015 Dec 8. PMID 26680107
- [Background] Haque MR, Ansari SH, Najmi AK, Ahmad MA. Monoterpene phenolic compound thymol prevents high fat diet induced obesity in murine model. Toxicol Mech Methods. 2014 Feb;24(2):116-23. doi: 10.3109/15376516.2013.861888. Epub 2013 Dec 5. PMID 24175857